CLINICAL TRIAL: NCT06546579
Title: Sensitivity of Self-collected Skin Sampling for Scabies: a Pilot Study
Acronym: SCRAPE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL86424.091.24
Record Dates: First submitted 2024-07-26; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies

STUDY DESIGN:
Intervention Model Description: The study design is cross-sectional in terms of the diagnostic process, which aims to determine the presence of scabies in an individual at a specific point in time. All participants will undergo the same diagnostic procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): All participants will be asked to perform self-sampling and irrespective of the result will receive current standard-of-care from their health care provider for their suspected scabies.
  Interventions: Diagnostic Test: Skin sampling

INTERVENTIONS:
Diagnostic Test: Skin sampling — All individuals will self-collect skin samples and swabs and fill in a questionnaire. Subsequently, all individuals will see a professional. The professional will collect skin samples and swabs as well.

SUMMARY:
In this cross-sectional diagnostic study, healthy adults aged 18 and older with suspected, clinical, or confirmed scabies will be recruited. The objective is to determine if the sensitivity of self-collected skin samples for scabies diagnosis is non-inferior to professional sampling, and compare the sensitivity and specificity of the polymerase chain reaction assay (PCR) versus microscopy.

DETAILED DESCRIPTION:
Scabies infestations have significantly increased globally in the last 10-20 years, including a threefold rise in the Netherlands over the past decade. Diagnosing scabies is challenging due to varied symptoms and low sensitivity of current microscopic methods. New diagnostic techniques like PCR, which offer higher sensitivity, are being investigated. The feasibility of self-collected skin samples is being explored to reduce the burden on healthcare services and address issues like autonomy, stigma, and privacy.

In this cross-sectional diagnostic study, healthy adults aged 18 and older with suspected, clinical, or confirmed scabies will be included. Primary endpoint is the sensitivity of self-collected versus professional skin samples for diagnosing scabies. Secondary endpoints include sensitivity of skin scrapings and swabs, and the sensitivity and specificity of PCR versus microscopy.

Participants will self-collect skin samples during a standard care visit. The process may be slightly sensitive but not painful. There are no direct benefits beyond standard care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have either suspected scabies, clinical scabies or confirmed scabies (see table 1)
* Providing informed consent (IC)

Exclusion Criteria:

* Individuals not speaking or understanding the Dutch or English language.
* Individuals who have been diagnosed with scabies in the last six weeks and had started treatment.
* Individuals who have used ivermectin for other diagnoses than scabies in the last six weeks.
* Individuals younger than 18 years.
* Individuals with immunosuppressive conditions (see appendix A).
* Any other condition, finding or situation which, in the opinion of the investigator, may significantly increase the risk to the individual because of participation in the study, affect the ability of the individual to participate in the study or impair interpretation of the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-08-21 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of self-collected skin samples for diagnosing scabies | through study completion, an average of one year
  The proportion of self-collected samples collected at the enrolment visit that are tested positive, divided by the total number of participants adjudged retrospectively to have had scabies at their enrolment visit, based on a composite clinical diagnosis.
The sensitivity of professionally-collected skin samples for diagnosing scabies | through study completion, an average of one year
  The proportion of professionally-collected samples collected at the enrolment visit that are tested positive, divided by the total number of participants adjudged retrospectively to have had scabies at their enrolment visit, based on a composite clinical diagnosis.

SECONDARY OUTCOMES:
The sensitivity of skin scrapings for diagnosing scabies | through study completion, an average of one year
  The proportion of skin scrapings at their enrolment visit (whether professionally or self-collected) that are tested positive by PCR, divided by the total number of participants adjudged retrospectively to have had scabies at baseline, based on a composite clinical diagnosis.
The sensitivity of skin swabs for diagnosing scabies | through study completion, an average of one year
  The proportion of skin swabs at their enrolment visit (whether professionally or self-collected) that are tested positive by PCR, divided by the total number of participants adjudged retrospectively to have had scabies at baseline, based on a composite clinical diagnosis.
The sensitivity and specificity of PCR on skin scraping for diagnosing active scabies infection | through study completion
  The proportion of participants adjudged to have had scabies at their enrolment visit (based on a retrospective composite clinical diagnosis), whose skin scraping at their enrolment visit (whether professionally or self-collected) are tested positive for scabies by PCR, and the proportion of participants adjudged retrospectively to have not had scabies at their enrolment visit whose skin scrapings are tested negative for scabies by PCR.
The sensitivity and specificity of microscopy on skin scraping for diagnosing active scabies infection | through study completion, an average of one year
  The proportion of participants adjudged to have had scabies at their enrolment visit (based on a retrospective composite clinical diagnosis), whose skin scraping at their enrolment visit (whether professionally or self-collected) are tested positive for scabies by microscopy, and the proportion of participants adjudged retrospectively to have not had scabies at their enrolment visit whose skin scrapings are tested negative* for scabies by microscopy.

OTHER OUTCOMES:
Proportion of participants whose self-sampling location is judged appropriate | through study completion, an average of one year
  Assessed by a professional at T=0 [adequate/non-adequate]
Motivation for self-collection of skin samples for scabies diagnostics | through study completion, an average of one year
  Motivation is assessed by items on the questionnaire related to the motivation for self-collection of skin samples for scabies diagnostics, along with the associated facilitators and barriers.
Demographic, clinical and epidemiological factors which influence the sensitivity of self-collected skin samples for scabies diagnosis. | through study completion, an average of one year
  Age, gender, highest level of education, signs/symptoms, living situation, skin color. source of transmission and transmission mode.

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No